CLINICAL TRIAL: NCT04131270
Title: Explaining Sedentary Behavior With the Revised Reflective + Impulsive Health Action Process Approach (HAPA) Model
Brief Title: Explaining Sedentary Behavior With Planning (the Revised HAPA Model)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Social Sciences and Humanities, Warsaw (Other)
Collaborators: National Science Centre, Poland (Other Government)
Responsible Party: Principal Investigator, Aleksandra Luszczynska, Professor of Psychology, University of Social Sciences and Humanities, Warsaw
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: USSHWarsaw; 2017/27/B/HS6/00092 (Other Grant/Funding Number: National Science Centre, Poland); 2021/43/O/HS6/00712/ (Other Grant/Funding Number: National Science Centre, Poland)
Record Dates: First submitted 2019-10-15; First posted 2019-10-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Sedentary Behavior
Keywords: Planning; Physical Activity
MeSH Terms: conditions — Sedentary Behavior; Motor Activity | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to an active control group (education on sedentary behavior and physical activity) or to a planning intervention (education on sedentary behavior and physical activity + education on how to form behavior change plans + forming a plan to change sedentary behavior using a planning sheet)
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Planning + Education (Experimental): 3 education sessions + 1 planning session (integrated into the 3rd education session); delivered face-to-face over 3 weeks (after the baseline measurement), individually.
  Planning: The planning materials and forms have sections: (a) instructions of what should be included in a good plan (the when, where, and how components), (b) formulating action and coping plans. Action plans (referring to when, when, and how the individual will act) as well as coping plans (referring to how to overcome potential difficulties) will be formed. After forming the plans individually, experimenters will discuss the plans with the participants.
  Interventions: Behavioral: Planning + Education; Behavioral: Education
- Education (Active Comparator): 3 education sessions; delivered face-to-face over 3 weeks (after the baseline measurement), individually.
  The education includes extended physical activity and sedentary behavior education using participant-educator discussions and printed materials.
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Planning + Education — Planning: Participants will fill in the planning forms that efer to replacing sedentary behavior with physical activity.
  The following behavior change techniques are included in the planning intervention protocol: action planning, barrier identification, prompting self-talk, relapse prevention/coping planning. Applications of all behavior change techniques would include references to planning.
  Arms: Planning + Education
Behavioral: Education — The education would include extended sedentary behavior and physical activity education, delivered face-to-face by the experimenters. The education includes: (1) the behavioral guidelines, tailored to age and health status of the participants, (2) the examples of exercises and their metabolic equivalent, and (3) the education about ways to break sedentary behavior with active breaks.

SUMMARY:
This study would investigate the effects of forming action plans on a reduction of sedentary behaviors. Participants will be randomly assigned to either active control group (education on sedentary behaviors and physical activity) or the intervention group (forming action plans referring to replacing sedentary activities with physical activity. The effects of the intervention will be evaluated at the 2-month follow-up and at the 8-month follow-up.

DETAILED DESCRIPTION:
The effects of three sessions (3 education sessions versus 3 education sessions+ forming plans to replace sedentary behavior with physical activity) will be investigated among participants from three age groups: adolescents (12-17 years old), adults (18-60 years old), and older adults (>60 years old). Compared to education only, forming plans about how to replace time spent on sedentary activities with physical activity is expected to result in a significantly larger change (a reduction) of sedentary time at the follow-up. Accelerometers will be used to evaluate short-term and mid-term changes in total sedentary time and the relative proportion of time spent on sedentary behavior vs light-intensity and moderate-to-vigorous- intensity physical activity.

Additionally, the study will observe changes in if the cognitions included in the Health Action Process Approach model (HAPA), such risk perception, self-efficacy, outcome expectancies, intention, action control, as well as changes in behavioral habit, presence of sedentary behavior cues in physical environment, and physical activity behavior. The observations will be conducted three times, at the baseline (before the intervention), the 2-month follow up, and at the 8-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* not meeting physical activity guidelines proposed by the World Health Organization

Exclusion Criteria:

* any existing diseases with contraindications for moderate intensity physical activity, confirmed by patient's primary care physician or a specialist in cardiovascular diseases/endocrinology/rehabilitation medicine providing care for the patient during the recruitment and follow-ups

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2020-01-02 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Sedentary behavior | change from the baseline sedentary behavior at 8 months
  minutes of sedentary behavior per day assessed with ActiGraph wGT3X-BT accelerometer

SECONDARY OUTCOMES:
The composition of waking time | change from the baseline composition of waking time at 8 months
  the proportion of time spent on sedentary behavior (minutes per day) to time spent on light-intensity physical activity (minutes per day) and moderate-to-vigorous physical activity (minutes per day) assessed with ActiGraph wGT3X-BT accelerometer
Physical activity | change from the baseline physical activity at 8 months
  minutes of light, moderate and vigorous intensity physical activity per day measured with ActiGraph wGT3X-BT accelerometer

OTHER OUTCOMES:
Sedentary behavior habit | change from the baseline sedentary behavior habit at 8 months
  Self-Reported Habit Scale; mean item score ranging from 1 to 4, higher scores indicate stronger sedentary behavior habit
Self-efficacy for reducing sedentary behavior | change from the baseline self-efficacy at 8 months
  9 self-efficacy questionnaire items; mean item score ranging from 1 to 4, higher scores indicate stronger self-efficacy
Risk perception | change from the baseline risk perception at 8 months
  3 questionnaire items to assess risk perception; mean item score ranging from 1 to 4, higher scores indicate higher risk perception
Outcome expectancies | change from the baseline outcome expectancies at 8 months
  18 items assessing positive (9 items) and negative (9 items) outcome expectancies; item score ranging from 1 to 4, higher scores indicate more positive outcome expectancies
Action control | change from the baseline outcome expectancies at 8 months
  10 questionnaire items assessing action control; mean item score ranging from 1 to 4, higher scores indicate stronger action control
Intention | change from the baseline intention at 8 months
  3 questionnaire items assessing intention to reduce sedentary behavior; mean item score ranging from 1 to 4, higher scores indicate stronger intention to reduce sedentary behavior
Self-reported planning | change from the baseline planning at 8 months
  4 questionnaire items assessing action planning; mean item score ranging from 1 to 4, higher scores indicate a higher level of self-reported planning
Environmental cues for sedentary behavior | change from the baseline planning at 8 months
  10 questionnaire items assessing physical environment cues for sedentary behavior and its reduction; the total sum score ranging from 0 to 10; higher scores indicate more environmental cues for sedentary behavior
Body mass index (BMI) | change from the baseline planning at 8 months
  Certified and standardized body weight scales (Beurer; European Union safety certificate; measurement error < 5%) and measuring rods will be used. Body mass index will be calculated using the following formula: body weight [in kg] divided by a square of body height (in meters). Body weight will be recorded in kilograms and body height will be recorded in meters.

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra Luszczynska, PhD, Principal Investigator — SWPS University of Social Sciences and Humanities
Locations (1):
- SWPS University of Social Sciences and Humanities, Wroclaw, Lower Silezia, Poland

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary, secondary, and additional outcome measures will be made available.
Supporting Information: Study Protocol, ICF
Time Frame: Respective data will be made available together with the submission of the manuscript reporting the findings for the main outcome (not later that within 2 years after the completion of data collection).
Access Criteria: Data will be uploaded on Open Science Framework, available to researchers who will have a respective link.

REFERENCES:
- [Background] Gardner B. A review and analysis of the use of 'habit' in understanding, predicting and influencing health-related behaviour. Health Psychol Rev. 2015;9(3):277-95. doi: 10.1080/17437199.2013.876238. Epub 2014 Jan 21. PMID 25207647
- [Background] Schwarzer R, Luszczynska A. Health action process approach. In: Norman P, Conner M, editors. Predicting and changing health behavior. Maidenead, UK: McGraw-Hill; 2015.
- [Background] Sallis JF, Spoon C, Cavill N, Engelberg JK, Gebel K, Parker M, Thornton CM, Lou D, Wilson AL, Cutter CL, Ding D. Co-benefits of designing communities for active living: an exploration of literature. Int J Behav Nutr Phys Act. 2015 Feb 28;12:30. doi: 10.1186/s12966-015-0188-2. PMID 25886356
- [Background] Maher JP, Conroy DE. A dual-process model of older adults' sedentary behavior. Health Psychol. 2016 Mar;35(3):262-72. doi: 10.1037/hea0000300. Epub 2015 Dec 21. PMID 26690644
- [Background] Keller C, Siegrist M. The weight management strategies inventory (WMSI). Development of a new measurement instrument, construct validation, and association with dieting success. Appetite. 2015 Sep;92:322-36. doi: 10.1016/j.appet.2015.05.037. Epub 2015 Jun 3. PMID 26048006
- [Background] Berli C, Loretini P, Radtke T, Hornung R, Scholz U. Predicting physical activity in adolescents: the role of compensatory health beliefs within the Health Action Process Approach. Psychol Health. 2014;29(4):458-74. doi: 10.1080/08870446.2013.865028. Epub 2013 Dec 20. PMID 24229317
- [Background] Luszczynska A, Hagger MS, Banik A, Horodyska K, Knoll N, Scholz U. Self-Efficacy, Planning, or a Combination of Both? A Longitudinal Experimental Study Comparing Effects of Three Interventions on Adolescents' Body Fat. PLoS One. 2016 Jul 13;11(7):e0159125. doi: 10.1371/journal.pone.0159125. eCollection 2016. PMID 27410961
- See also: Study protocol in Polish — https://drive.google.com/a/swps.edu.pl/file/d/1zP8QcSXBCtew5yugMEi47DriT_1uxtv2/view?usp=sharing